CLINICAL TRIAL: NCT01762280
Title: A Phase I Study of Famitinib Malate in Patients With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other); Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTN-I
Record Dates: First submitted 2012-12-26; First posted 2013-01-07 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2013-01

CONDITIONS: Advanced Solid Tumor
Keywords: Famitinib; Advanced Solid tumor; Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Famitinib Malate (Experimental): Famitinib either at 4,8,13,20,27,36 mg, p.o. once daily
  Interventions: Drug: Famitinib Malate Capsule

INTERVENTIONS:
Drug: Famitinib Malate Capsule

SUMMARY:
Famitinib is a novel oral multitargeted tyrosine kinase inhibitor with antitumor and antiangiogenic activities. This study is designed to evaluate the safety and tolerability of Famitinib in patients with solid tumor

DETAILED DESCRIPTION:
1. To evaluate the safety and tolerability of Famitinib, and the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT).
2. To determine the pharmacokinetic profile of Famitinib and its metabolites .
3. To assess preliminary antitumor activity .
4. To determine preliminary dose and regimen for phase II study .

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed advanced or metastatic solid tumor，at least one measurable lesion, larger than 10 mm in diameter by spiral CT scan(scanning layer ≤ 5 mm )
* no standard therapy protocol available according to patients'condition
* both sex, age 18 to 65
* ECOG 0-1
* Life expectancy more than 3 months
* ALT,AST,TB≤1.5(UNL),normal serum creatinine level, normal electrolyte or can be corrected by medication
* Subjects receiving damage caused by other therapeutic has been restored, the interval more than six weeks since the last receiving nitroso or mitomycin; more than 4 weeks since last receiving radiotherapy, other cytotoxic drugs or surgery
* Understand and agree to sign informed consent form.

Exclusion Criteria:

* Peripheral neuropathy ≥ Grade 2(according to NCI-CTC 3.0)
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg by using single agent therapy, >Grade 1 (NCI-CTCAE 3.0 ) myocardial ischemia, arrhythmia,cardiac function insufficiency
* PT, APTT, TT, Fbg abnormal(PT>16s,APTT>43s,TT>21s,Fbg<2g/L), or have hemorrhagic tendency or receiving the therapy of thrombolysis or anticoagulation
* Active peptic ulcer
* Previously medication include sunitinib
* More than 4 weeks since the last clinical trial
* Pregnant or lactating women
* Women of childbearing age do not take effective contraceptive measures
* Allergies, or known allergy history to components of the drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) | 2 months
Dose-limiting toxicity(DLT) | 2 months

SECONDARY OUTCOMES:
Pharmacokinetics | 2 months
  Famitinib pharmacokinetic parameters , include AUC, Cmax, Tmax, and t1/2
Objective response rate | 2 months
Number of volunteers with adverse events | 2 months
Pharmacodynamics | 2 months
  The response of Famitinib on tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, M.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Dafang Zhong, Ph.D, Principal Investigator — Chinese Academy of Science Shanghai Institution of Materia Medica
Locations (1):
- Cancer Institute and Hospital Chinese Academy of Medical Sciences, Beijing, China